## PROTOCOL NUMBER CMS-005 PHASE I STUDY OF AD5 [E1-, E2B-]-HER2/NEU VACCINE (ETBX-021) IN SUBJECTS WITH UNRESECTABLE LOCALLY ADVANCED OR METASTATIC HER2-EXPRESSING BREAST CANCER

| IND Number: | 016,871 |
|---|---|
| Principal Investigator: | Hatem Soliman, MD |
| | Moffitt Cancer Center |
| | 12902 Magnolia Drive |
| | Tampa, Florida 33612 |
| | Email: hatem.soliman@moffitt.org |
| | Office Phone: 813-745-4933 |
| Clinical Study Sponsor: | NantBioScience, Inc. |
| Sponsor Contact: | Wayne R. Godfrey, MD |
| (For medical questions/emergencies) | Chief Medical Officer |
| | Medical and Safety Monitor |
| | Email: wayne@etubics.com |
| | Office Phone: 206-838-5110, Ext 9 |
| | Mobile Phone: 650-521-2770 |
| Sponsor Contact: | Jackie Imm, BA |
| (For study administration, operations, and | Clinical Trial Manager |
| execution questions) | Email: Jackie.Imm@NantBio.com |
| • | Office Phone: 919-694-6315 |
| SAE Reporting: | Submit SAE Reports to one (1) of the |
| | following: |
| | SAE Email: SAE.Reporting@NantBio.com |
| | Fax: 800-853-3497 |

| Protocol Version | Date |
|---------------------------|------------------|
| Original Protocol CMS-005 | 26 February 2016 |

ETBX-021 Clinical Trial Protocol: CMS-005

### PROTOCOL SYNOPSIS

### Name of Sponsor/Company:

NantBioScience, Inc.

### Name of Investigational Product:

Ad5 [E1-, E2b-]-HER2/neu Vaccine, Suspension for Injection (ETBX-021)

### **Name of Active Ingredient:**

Ad5 [E1-, E2b-]-HER2/neu

### **Title of Study:**

Phase I Study of Ad5 [E1-, E2b-]-HER2/neu Vaccine (ETBX-021) in Subjects with Unresectable Locally Advanced or Metastatic HER2-Expressing Breast Cancer

### **Study Number:**

CMS-005

### **Study Phase:**

Phase I

### **Primary Objectives:**

• Determine the overall safety and recommended phase 2 dose of ETBX-021 when administered subcutaneously (SC) every 3 weeks for three injections followed by three booster injections at 3-month intervals to subjects with HER2-expressing breast cancer.

### **Secondary Objectives:**

• Make preliminary assessments of objective response rate (ORR), disease control rate (DCR), duration of response, progression-free survival (PFS), and overall survival (OS) in subjects with HER2-expressing breast cancer treated with ETBX-021.

### **Exploratory Objectives:**

Evaluate the immunogenicity of ETBX-021 and determine the genomic and proteomic profile
of subjects' tumors to identify gene mutations, gene amplifications, RNA-expression levels,
and protein-expression levels. Correlations between genomic/proteomic profiles and efficacy
outcomes will be assessed.

### **Primary Endpoints:**

- Dose-limiting toxicities (DLTs) and maximum tolerated dose (MTD) or highest tested dose (HTD).
- Treatment-emergent adverse event (AEs) and serious adverse events (SAEs).
- Clinically significant changes in safety laboratory tests, physical examinations, electrocardiograms (ECGs), left ventricular ejection fraction (LVEF), and vital signs.

### **Secondary Endpoints:**

- ORR (confirmed complete or partial response) according to the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
- DCR (confirmed response or stable disease lasting for at least 6 months).
- Duration of response.
- PFS.
- OS.

### **Exploratory** Endpoints:

- Immunogenicity of ETBX-021 by flow cytometric analysis of T-cell frequency, activation status, cytokine profiles, and antibody levels.
- Genetic and proteomic profiling and correlates with efficacy.

### **Study Design:**

This is a Phase I trial in subjects with unresectable locally advanced or metastatic HER2-low expressing (IHC 1+ or 2+) breast cancer. The study will be conducted in two parts: the first part will involve dose escalation using a 3 + 3 design, and the second part will involve the expansion of the MTD or HTD to further evaluate safety, preliminary efficacy, and immunogenicity. In the first part, 3 to 6 subjects will be sequentially enrolled starting at dose cohort 1. Subjects will be assessed for dose-limiting toxicities (DLTs).

- Cohort 1: 5 x 10<sup>10</sup> virus particles (VP).
- Cohort 2: 5 x 10<sup>11</sup> VP.
- If needed, dose de-escalation cohort (cohort -1): 5 x 10<sup>9</sup> VP.

Dose expansion will occur when the MTD or HTD has been determined. An additional 12 subjects will be enrolled in the dose expansion component of the trial, for a total of 18 subjects at the MTD or HTD.

### **Enrollment (planned):**

Up to 30 subjects will be enrolled in the study. In the dose escalation component, 3 to 6 subjects will be sequentially enrolled starting at Cohort 1. In the dose expansion component (i.e., once the MTD or HTD has been identified), an additional 12 subjects will be enrolled for a total of 18 subjects in the MTD/HTD cohort to obtain further safety, preliminary efficacy, and immunogenicity data.

### **Diagnosis and Main Criteria for Inclusion:**

Subjects must have histologically confirmed unresectable locally advanced or metastatic breast cancer that expresses HER2 (IHC 1+ or 2+). Subjects with HER2 IHC 3+ tumors are excluded.

### **Investigational Product, Dosage, and Mode of Administration:**

ETBX-021 (5 x 10<sup>9</sup>, 5 x 10<sup>10</sup>, or 5 x 10<sup>11</sup> VP in 1.0 mL) will be administered by SC injection every 3 weeks for 3 injections, followed by 3 booster injections at 3-month intervals.

### **Duration of Treatment:**

Subjects will receive treatment for up to 42 weeks (injections at 0, 3, and 6 weeks with booster injections at 18, 30, and 42 weeks) or until they experience progressive disease or unacceptable toxicity, withdraw consent, or if the Investigator feels it is no longer in their best interest to continue treatment.

### Reference Therapy, Dosage, and Mode of Administration:

Not applicable.

### **Criteria for Evaluation:**

**Safety:** Safety endpoints include assessments of DLT, MTD or HTD, treatment-emergent AEs, SAEs, and clinically significant changes in safety laboratory tests, physical examinations, ECGs, LVEF, and vital signs. Toxicities will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03.

**Efficacy:** Tumor response (ORR and DCR) will be evaluated according to RECIST Version 1.1; duration of response, PFS, and OS will also be evaluated.

**Exploratory Immune Analysis:** Immune responses will be detected and quantified in flow cytometry-based and serum assays.

Clinical Trial Protocol: CMS-005

**Exploratory Molecular Profiling and Analysis:** Genomic sequencing of tumor cells relative to non-tumor cells to identify the genomic variances that may contribute to response or disease progression and provide an understanding of molecular abnormalities; RNA sequencing to provide expression data and give relevance to DNA mutations; and quantitative proteomics to determine the exact amounts of specific proteins and to confirm expression of genes predictive of response and disease progression.

### **Statistical Methods:**

The rate of DLTs and the MTD or HTD will be assessed. Overall safety will be assessed by descriptive analyses using tabulated frequencies of AEs by grade using CTCAE Version 4.03 within dose cohorts and for the overall study population in terms of treatment-emergent AEs, SAEs, and clinically significant changes in safety laboratory tests, physical examinations, ECGs, LVEF, and vital signs. ORR and DCR will be evaluated according to RECIST Version 1.1 by dose cohort and overall; duration of response will also be evaluated. PFS and OS will be analyzed using Kaplan-Meier methods by dose cohort and overall.

ETBX-021
Clinical Trial Protocol: CMS-005
NantBioScience, Inc.

Figure 1: Study Design and Treatment Schema



ETBX-021 NantBioScience, Inc.

Clinical Trial Protocol: CMS-005

**Table 3:** Time and Events Schedule

| Assessment | Screening | Baseline | (Eve | Treatment Boosters (Every 3-Week Dosing) (Every 3-Month Dosing) | | | | | | End of<br>Study | Post<br>Study<br>Follow<br>Up | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | Day -28 to -7 | Day<br>-7 to 1 | 0 | 3 | 6 | 9 | 18 | 21 | 30 | 33 | 42 | 45 | |
| Clinic Visit | X | X | X | X | X | X | X | | X | | X | | X |
| Informed Consent | X | | | | | | | | | | | | |
| Inclusion/Exclusion | X | X | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | |
| Physical Examination, Height <sup>a</sup> ,<br>Weight, ECOG | X | X | X | X | X | X | X | | X | | X | | X |
| Medical History <sup>b</sup> | X | X | | | | | | | | | | | |
| Confirm HER2 Expression | X | | | | | | | | | | | | |
| Concomitant Medications | X | X | X | X | X | X | X | | X | | X | | X |
| Vital Signs <sup>c</sup> | X | X | X | X | X | X | X | | X | | X | | X |
| 12-Lead ECG | X | | | | | X | X | | X | | X | | X |
| Echocardiogram/MUGA <sup>d</sup> | X | | | | | X | X | | X | | X | | X |
| Confirm Contraceptive Measures <sup>e</sup> | X | | | | | | | | | | | | |
| Study Drug Injection/ Injection<br>Site Reaction Monitoring <sup>f</sup> | | | X | X | X | | X | | X | | X | | |
| Dispensation of Subject Diary<br>Card <sup>g</sup> | | | X | X | X | | X | | X | | X | | |
| Review of Subject Diary Card <sup>g</sup> | | | | X | X | X | | X | | X | | X | |

| Assessment | Screening | Baseline | (Eve | Treatment Boosters (Every 3-Week Dosing) (Every 3-Month Dosing) | | | | | | End of<br>Study | Post<br>Study<br>Follow<br>Up | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | Day<br>-28 to -7 | Day<br>-7 to 1 | 0 | 3 | 6 | 9 | 18 | 21 | 30 | 33 | 42 | 45 | | |
| Telephone Contact 72 Hours Post<br>Injection | | | X | X | X | | X | | X | | X | | | |
| Tumor Imaging <sup>h</sup> | | X | | | | X | | X | | X | | X | X | |
| Pregnancy Test <sup>i</sup> | X | | X | X | X | | X | | X | | X | | X | |
| Urinalysis | X | | | | | X | | | X | | | | X | |
| Chemistry Panel | X | X | X | X | X | X | X | | X | | X | | X | |
| CBC, Differential, Platelets | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Coagulation | X | | | | | X | | | | | X | | X | |
| Serum Virology (HIV, HBV, HCV) | X | | | | | | | | | | | | | |
| Adverse Events | | X | X | X | X | X | X | X | X | X | X | X | X | |
| Exploratory Immune Analysis | | X | X | X | X | X | X | X | X | X | X | X | | |
| Exploratory Genomics and<br>Proteomics Molecular Analysis | | X | | | | | | | | | | | | |
| Telephone Follow Up <sup>j</sup> | | | | | | | | | | | | | | X |

Clinical Trial Protocol: CMS-005

### APPENDIX 2. SPONSOR SIGNATURE

| Study Title: | Phase I Study of Ad5 [E1-, E2b-]-HER2/neu Vaccine (ETBX-021) in Subjects with Unresectable Locally Advanced or Metastatic HER2-Expressing Breast Cancer |
|---|---|
| Study Number: | CMS-005 |
| Final Date: | 26 February 2016 |

This clinical study protocol was subject to critical review and has been approved by the Sponsor. The following personnel contributed to writing and/or approving this protocol:

Signed:

Wayne R. Godfrey, MD Chief Medical Officer Medical and Safety Monitor NantBioScience, Inc.

### PROTOCOL NUMBER CMS-005 PHASE I STUDY OF AD5 [E1-, E2B-]-HER2/NEU VACCINE (ETBX-021) IN SUBJECTS WITH

### UNRESECTABLE LOCALLY ADVANCED OR METASTATIC HER2-EXPRESSING BREAST CANCER

| IND Number: | 016,871 |
|---|---|
| Principal Investigator: | Hatem Soliman, MD |
| | Moffitt Cancer Center |
| | 12902 Magnolia Drive |
| | Tampa, Florida 33612 |
| | Email: hatem.soliman@moffitt.org |
| | Office Phone: 813-745-4933 |
| Clinical Study Sponsor: | NantBioScience, Inc. |
| Sponsor Contact: | Wayne R. Godfrey, MD |
| (For medical questions/emergencies) | Chief Medical Officer |
| | Medical and Safety Monitor |
| | Email: wayne@etubics.com |
| | Office Phone: 206-838-5110, Ext 9 |
| | Mobile Phone: 650-521-2770 |
| Sponsor Contact: | Jackie Imm, BA |
| (For study administration, operations, and | Clinical Trial Manager |
| execution questions) | Email: Jackie.Imm@NantBio.com |
| - | Office Phone: 919-694-6315 |
| SAE Reporting: | Submit SAE Reports to one (1) of the |
| <del>-</del> - | following: |
| | SAE Email: SAE.Reporting@NantBio.com |
| | Fax: 800-853-3497 |

| Protocol Version | Date |
|------------------------------|------------------|
| Original Protocol CMS-005 | 26 February 2016 |
| Protocol CMS-005 Amendment 1 | 21 April 2016 |

### PROTOCOL SYNOPSIS

### Name of Sponsor/Company:

NantBioScience, Inc.

ETBX-021

### **Name of Investigational Product:**

Ad5 [E1-, E2b-]-HER2/neu Vaccine, Suspension for Injection (ETBX-021)

### Name of Active Ingredient:

Ad5 [E1-, E2b-]-HER2/neu

### Title of Study:

Phase I Study of Ad5 [E1-, E2b-]-HER2/neu Vaccine (ETBX-021) in Subjects with Unresectable Locally Advanced or Metastatic HER2-Expressing Breast Cancer

### **Study Number:**

CMS-005

### **Study Phase:**

Phase I

### **Primary Objectives:**

• Determine the overall safety and recommended phase 2 dose of ETBX-021 when administered subcutaneously (SC) every 3 weeks for three injections followed by three booster injections at 3-month intervals to subjects with HER2-expressing breast cancer.

### **Secondary Objectives:**

• Make preliminary assessments of objective response rate (ORR), disease control rate (DCR), duration of response, progression-free survival (PFS), and overall survival (OS) in subjects with HER2-expressing breast cancer treated with ETBX-021.

### **Exploratory Objectives:**

• Evaluate the immunogenicity of ETBX-021 and determine the genomic and proteomic profile of subjects' tumors to identify gene mutations, gene amplifications, RNA-expression levels, and protein-expression levels. Correlations between genomic/proteomic profiles and efficacy outcomes will be assessed.

### **Primary Endpoints:**

- Dose-limiting toxicities (DLTs) and maximum tolerated dose (MTD) or highest tested dose (HTD).
- Treatment-emergent adverse event (AEs) and serious adverse events (SAEs).
- Clinically significant changes in safety laboratory tests, physical examinations, electrocardiograms (ECGs), left ventricular ejection fraction (LVEF), and vital signs.

### **Secondary Endpoints:**

- ORR (confirmed complete or partial response) according to the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
- DCR (confirmed response or stable disease lasting for at least 6 months).
- Duration of response.
- PFS.

Clinical Trial Protocol: CMS-005 Amendment 1

• OS.

### **Exploratory Endpoints:**

- Immunogenicity of ETBX-021 by flow cytometric analysis of T-cell frequency, activation status, cytokine profiles, and antibody levels.
- Genetic and proteomic profiling and correlations with efficacy.

### **Study Design:**

This is a Phase I trial in subjects with unresectable locally advanced or metastatic HER2-low expressing (IHC 1+ or 2+) breast cancer. The study will be conducted in two parts: the first part will involve dose escalation using a 3 + 3 design, and the second part will involve the expansion of the MTD or HTD to further evaluate safety, preliminary efficacy, and immunogenicity. In the first part, 3 to 6 subjects will be sequentially enrolled starting at dose cohort 1. Subjects will be assessed for dose-limiting toxicities (DLTs).

- Cohort 1: 5 x 10<sup>10</sup> virus particles (VP).
- Cohort 2: 5 x 10<sup>11</sup> VP.
- If needed, dose de-escalation cohort (cohort -1): 5 x 10<sup>9</sup> VP.

Dose expansion will occur when the MTD or HTD has been determined. An additional 12 subjects will be enrolled in the dose expansion component of the trial, for a total of 18 subjects at the MTD or HTD.

### **Enrollment (planned):**

Up to 30 subjects will be enrolled in the study. In the dose escalation component, 3 to 6 subjects will be sequentially enrolled starting at Cohort 1. In the dose expansion component (i.e., once the MTD or HTD has been identified), an additional 12 subjects will be enrolled for a total of 18 subjects in the MTD/HTD cohort to obtain further safety, preliminary efficacy, and immunogenicity data.

### Diagnosis and Main Criteria for Inclusion:

Subjects must have histologically confirmed unresectable locally advanced or metastatic breast cancer that expresses HER2 (IHC 1+ or 2+). Subjects with HER2 IHC 3+ tumors are excluded.

### **Investigational Product, Dosage, and Mode of Administration:**

ETBX-021 (5 x 10<sup>9</sup>, 5 x 10<sup>10</sup>, or 5 x 10<sup>11</sup> VP in 1.0 mL) will be administered by SC injection every 3 weeks for 3 injections, followed by 3 booster injections at 3-month intervals.

### **Duration of Treatment:**

Subjects will receive treatment for up to 42 weeks (injections at 0, 3, and 6 weeks with booster injections at 18, 30, and 42 weeks) or until they experience progressive disease or unacceptable toxicity, withdraw consent, or if the Investigator feels it is no longer in their best interest to continue treatment.

### Reference Therapy, Dosage, and Mode of Administration:

Not applicable.

### **Criteria for Evaluation:**

**Safety:** Safety endpoints include assessments of DLT, MTD or HTD, treatment-emergent AEs, SAEs, and clinically significant changes in safety laboratory tests, physical examinations, ECGs, LVEF, and vital signs. Toxicities will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03.

**Efficacy:** Tumor response (ORR and DCR) will be evaluated according to RECIST Version 1.1; duration of response, PFS, and OS will also be evaluated.

Clinical Trial Protocol: CMS-005 Amendment 1

**Exploratory Immune Analysis:** Immune responses will be detected and quantified in flow cytometry-based and serum assays.

Exploratory Molecular Profiling and Analysis and its Rationale: Genomic sequencing of tumor cells from tissue relative to non-tumor cells from whole blood will be profiled to identify the genomic variances that may contribute to response or disease progression and provide an understanding of molecular abnormalities. RNA sequencing will be conducted to provide expression data and give relevance to DNA mutations. Quantitative proteomics analysis will be conducted to determine the exact amounts of specific proteins and to confirm expression of genes that are correlative of response to vaccine immunotherapy and disease progression. All genomic, transcriptomic, and proteomic molecular analyses will be retrospective and exploratory.

### **Statistical Methods:**

The rate of DLTs and the MTD or HTD will be assessed. Overall safety will be assessed by descriptive analyses using tabulated frequencies of AEs by grade using CTCAE Version 4.03 within dose cohorts and for the overall study population in terms of treatment-emergent AEs, SAEs, and clinically significant changes in safety laboratory tests, physical examinations, ECGs, LVEF, and vital signs. ORR and DCR will be evaluated according to RECIST Version 1.1 by dose cohort and overall; duration of response will also be evaluated. PFS and OS will be analyzed using Kaplan-Meier methods by dose cohort and overall.

Figure 1: Study Design and Treatment Schema



ETBX-021 NantBioScience, Inc.

Clinical Trial Protocol: CMS-005 Amendment 1

**Table 3:** Time and Events Schedule

| Assessment | Screening | | Treatment Boosters (Every 3-Week Dosing) (Every 3-Month Dosing) | | | | | | | End<br>of<br>Study | Post<br>Study<br>Follow<br>Up | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | Day<br>-28 to -1 | Baseline/ | 3 | 6 | 9 | 18 | 21 | 30 | 33 | 42 | 45 | |
| Clinic Visit | X | X | X | X | X | X | X | X | X | X | X | X |
| Informed Consent | X | | | | | | | | | | | |
| Inclusion/Exclusion | X | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | |
| Physical Examination, Height <sup>a</sup> ,<br>Weight, ECOG | X <sup>b</sup> | $X^{b}$ | X | X | X | X | | X | | X | | X |
| Medical History <sup>c</sup> | X | X | | | | | | | | | | |
| Confirm HER2 Expression <sup>d</sup> | X | | | | | | | | | | | |
| Concomitant Medications | X | X | X | X | X | X | | X | | X | | X |
| Vital Signs <sup>e</sup> | X | X | X | X | X | X | | X | | X | | X |
| 12-Lead ECG | X | | | | X | X | | X | | X | | X |
| Echocardiogram/MUGA <sup>f</sup> | X | | | | X | X | | X | | X | | X |
| Confirm Contraceptive Measures <sup>g</sup> | X | | | | | | | | | | | |
| Study Drug Injection/ Injection<br>Site Reaction Monitoring <sup>h</sup> | | X | X | X | | X | | X | | X | | |
| Dispensation of Subject Diary<br>Card <sup>i</sup> | | X | X | X | | X | | X | | X | | |

ETBX-021 Clinical Trial Protocol: CMS-005 Amendment 1

| Assessment | Screening | | Treatment Boosters (Every 3-Week Dosing) (Every 3-Month Dosing) | | | | | | End<br>of<br>Study | Post<br>Study<br>Follow<br>Up | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | Day<br>-28 to -1 | Baseline/ | 3 | 6 | 9 | 18 | 21 | 30 | 33 | 42 | 45 | | |
| Review of Subject Diary Card <sup>i</sup> | | | X | X | X | | X | | X | | X | X | |
| Telephone Contact 72 Hours Post<br>Injection | | X | X | X | | X | | X | | X | | | |
| Tumor Imaging <sup>j</sup> | X | | | | X | X | | X | | X | | X | |
| Pregnancy Test <sup>k</sup> | X <sup>b</sup> | X <sup>b</sup> | X | X | | X | | X | | X | | X | |
| Urinalysis | X | | | | X | | | X | | | | X | |
| Chemistry Panel | X <sup>b</sup> | X <sup>b</sup> | X | X | X | X | | X | | X | | X | |
| CBC, Differential, Platelets | X <sup>b</sup> | X <sup>b</sup> | X | X | X | X | | X | | X | | X | |
| Coagulation | X | | | | X | | | | | X | | X | |
| Serum Virology (HIV, HBV, HCV) <sup>l</sup> | X | | | | | | | | | | | | |
| Adverse Events | | X | X | X | X | X | X | X | X | X | X | X | |
| Exploratory Immune Analysis | | X | X | X | X | X | X | X | X | X | X | | |
| Exploratory Genomics and<br>Proteomics Molecular Analysis | X | | | | | | | | | | | | |
| Telephone Follow Up <sup>m</sup> | | _ | | | | | | | | | | | X |

### APPENDIX 2. SPONSOR SIGNATURE

| Study Title: | Phase I Study of Ad5 [E1-, E2b-]-HER2/neu Vaccine (ETBX-021) in Subjects with Unresectable Locally Advanced or Metastatic HER2-Expressing Breast Cancer |
|---|---|
| Study Number: | CMS-005, Amendment 1 |
| Final Date: | 21 April 2016 |

This clinical study protocol was subject to critical review and has been approved by the Sponsor. The following personnel contributed to writing and/or approving this protocol:

Signed:

Wayne R. Godfrey, MD Chief Medical Officer

Medical and Safety Monitor

NantBioScience, Inc.

### PROTOCOL NUMBER CMS-005

### PHASE I STUDY OF AD5 [E1-, E2B-]-HER2/NEU VACCINE (ETBX-021) IN SUBJECTS WITH UNRESECTABLE LOCALLY ADVANCED OR METASTATIC HER2-LOW-EXPRESSING (IHC 1+/2+) BREAST CANCER

| IND Number: | 016,871 |
|---|---|
| Principal Investigator: | Hatem Soliman, MD |
| | Moffitt Cancer Center |
| | 12902 Magnolia Drive |
| | Tampa, Florida 33612 |
| | Email: hatem.soliman@moffitt.org |
| | Office Phone: 813-745-4933 |
| Clinical Study Sponsor: | NantBioScience, Inc. |
| Sponsor Contact: | Wayne R. Godfrey, MD |
| (For medical questions/emergencies) | Chief Medical Officer |
| | Medical and Safety Monitor |
| | Email: wayne@etubics.com |
| | Office Phone: 206-838-5110, Ext 9 |
| | Mobile Phone: 650-521-2770 |
| <b>Sponsor Contact:</b> | Jackie Imm, BA |
| (For study administration, operations, and | Clinical Trial Manager |
| execution questions) | Email: Jackie.Imm@NantBio.com |
| | Office Phone: 919-694-6315 |
| SAE Reporting: | Submit SAE Reports to one (1) of the |
| | following: |
| | SAE Email: SAE.Reporting@NantBio.com |
| | Fax: 800-853-3497 |

| Protocol Version | Date |
|------------------------------|------------------|
| Original Protocol CMS-005 | 26 February 2016 |
| Protocol CMS-005 Amendment 1 | 20 April 2016 |
| Protocol CMS-005 Amendment 2 | 25 May 2016 |

### PROTOCOL SYNOPSIS

### Name of Sponsor/Company:

NantBioScience, Inc.

### **Name of Investigational Product:**

Ad5 [E1-, E2b-]-HER2/neu Vaccine, Suspension for Injection (ETBX-021)

### Name of Active Ingredient:

Ad5 [E1-, E2b-]-HER2/neu

### Title of Study:

Phase I Study of Ad5 [E1-, E2b-]-HER2/neu Vaccine (ETBX-021) in Subjects with Unresectable Locally Advanced or Metastatic HER2-Low-Expressing (IHC 1+/2+) Breast Cancer

### **Study Number:**

CMS-005

### **Study Phase:**

Phase I

### **Primary Objectives:**

• Determine the overall safety and recommended phase 2 dose of ETBX-021 when administered subcutaneously (SC) every 3 weeks for three injections followed by three booster injections at 3-month intervals to subjects with HER2-low-expressing breast cancer.

### **Secondary Objectives:**

 Make preliminary assessments of objective response rate (ORR), disease control rate (DCR), duration of response, progression-free survival (PFS), and overall survival (OS) in subjects with HER2-low-expressing breast cancer treated with ETBX-021.

### **Exploratory Objectives:**

• Evaluate the immunogenicity of ETBX-021 and determine the genomic and proteomic profile of subjects' tumors to identify gene mutations, gene amplifications, RNA-expression levels, and protein-expression levels. Correlations between genomic/proteomic profiles and efficacy outcomes will be assessed.

### **Primary Endpoints:**

- Dose-limiting toxicities (DLTs) and maximum tolerated dose (MTD) or highest tested dose (HTD).
- Treatment-emergent adverse event (AEs) and serious adverse events (SAEs).
- Clinically significant changes in safety laboratory tests, physical examinations, electrocardiograms (ECGs), left ventricular ejection fraction (LVEF), and vital signs.

### **Secondary Endpoints:**

- ORR (confirmed complete or partial response) according to the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
- DCR (confirmed response or stable disease lasting for at least 6 months).
- Duration of response.
- PFS.

Clinical Trial Protocol: CMS-005 Amendment 2

• OS.

### **Exploratory Endpoints:**

- Immunogenicity of ETBX-021 by flow cytometric analysis of T-cell frequency, activation status, cytokine profiles, and antibody levels.
- Genetic and proteomic profiling and correlations with efficacy.

### **Study Design:**

This is a Phase I trial in subjects with unresectable locally advanced or metastatic HER2-low-expressing (IHC 1+ or 2+) breast cancer. The study will be conducted in two parts: the first part will involve dose escalation using a 3 + 3 design, and the second part will involve the expansion of the MTD or HTD to further evaluate safety, preliminary efficacy, and immunogenicity. In the first part, 3 to 6 subjects will be sequentially enrolled starting at dose cohort 1. Subjects will be assessed for dose-limiting toxicities (DLTs).

- Cohort 1: 5 x 10<sup>10</sup> virus particles (VP).
- Cohort 2: 5 x 10<sup>11</sup> VP.
- If needed, dose de-escalation cohort (cohort -1): 5 x 10<sup>9</sup> VP.

Dose expansion will occur when the MTD or HTD has been determined. An additional 12 subjects will be enrolled in the dose expansion component of the trial, for a total of 18 subjects at the MTD or HTD.

### **Enrollment (planned):**

Up to 30 subjects will be enrolled in the study. In the dose escalation component, 3 to 6 subjects will be sequentially enrolled starting at Cohort 1. In the dose expansion component (i.e., once the MTD or HTD has been identified), an additional 12 subjects will be enrolled for a total of 18 subjects in the MTD/HTD cohort to obtain further safety, preliminary efficacy, and immunogenicity data.

### **Diagnosis and Main Criteria for Inclusion:**

Subjects must have histologically confirmed unresectable locally advanced or metastatic breast cancer that expresses HER2 (IHC 1+ or 2+). Subjects with HER2 IHC 3+ tumors are excluded.

### **Investigational Product, Dosage, and Mode of Administration:**

ETBX-021 (5 x  $10^9$ , 5 x  $10^{10}$ , or 5 x  $10^{11}$  VP in 1.0 mL) will be administered by SC injection every 3 weeks for 3 injections, followed by 3 booster injections at 3-month intervals.

### **Duration of Treatment:**

Subjects will receive treatment for up to 42 weeks (injections at 0, 3, and 6 weeks with booster injections at 18, 30, and 42 weeks) or until they experience progressive disease or unacceptable toxicity, withdraw consent, or if the Investigator feels it is no longer in their best interest to continue treatment.

### Reference Therapy, Dosage, and Mode of Administration:

Not applicable.

### **Criteria for Evaluation:**

**Safety:** Safety endpoints include assessments of DLT, MTD or HTD, treatment-emergent AEs, SAEs, and clinically significant changes in safety laboratory tests, physical examinations, ECGs, LVEF, and vital signs. Toxicities will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03.

**Efficacy:** Tumor response (ORR and DCR) will be evaluated according to RECIST Version 1.1; duration of response, PFS, and OS will also be evaluated.

Clinical Trial Protocol: CMS-005 Amendment 2

**Exploratory Immune Analysis:** Immune responses will be detected and quantified in flow cytometry-based and serum assays.

Exploratory Molecular Profiling and Analysis and its Rationale: Genomic sequencing of tumor cells from tissue relative to non-tumor cells from whole blood will be profiled to identify the genomic variances that may contribute to response or disease progression and provide an understanding of molecular abnormalities. RNA sequencing will be conducted to provide expression data and give relevance to DNA mutations. Quantitative proteomics analysis will be conducted to determine the exact amounts of specific proteins and to confirm expression of genes that are correlative of response to vaccine immunotherapy and disease progression. All genomic, transcriptomic, and proteomic molecular analyses will be retrospective and exploratory.

### **Statistical Methods:**

The rate of DLTs and the MTD or HTD will be assessed. Overall safety will be assessed by descriptive analyses using tabulated frequencies of AEs by grade using CTCAE Version 4.03 within dose cohorts and for the overall study population in terms of treatment-emergent AEs, SAEs, and clinically significant changes in safety laboratory tests, physical examinations, ECGs, LVEF, and vital signs. ORR and DCR will be evaluated according to RECIST Version 1.1 by dose cohort and overall; duration of response will also be evaluated. PFS and OS will be analyzed using Kaplan-Meier methods by dose cohort and overall.

Figure 1: Study Design and Treatment Schema



ETBX-021 NantBioScience, Inc.

Clinical Trial Protocol: CMS-005 Amendment 2

**Table 3:** Time and Events Schedule

| Assessment | Screening | | Treatment Boosters (Every 3-Week Dosing) (Every 3-Month Dosing) | | | | | | | | | End<br>of<br>Study | Post<br>Study<br>Follow<br>Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | Day -28 to -1 | Baseline/ | 3 | 6 | 9 | 18 | 21 | 30 | 33 | 42 | 45 | | |
| Clinic Visit | X | X | X | X | X | X | X | X | X | X | X | X | |
| Informed Consent | X | | | | | | | | | | | | |
| Inclusion/Exclusion | X | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | |
| Physical Examination, Height <sup>a</sup> , Weight, ECOG | X <sup>b</sup> | $X^b$ | X | X | X | X | | X | | X | | X | |
| Medical History <sup>c</sup> | X | X | | | | | | | | | | | |
| Confirm HER2 Expression <sup>d</sup> | X | | | | | | | | | | | | |
| Concomitant Medications | X | X | X | X | X | X | | X | | X | | X | |
| Vital Signs <sup>e</sup> | X | X | X | X | X | X | | X | | X | | X | |
| 12-Lead ECG | X | | | | X | X | | X | | X | | X | |
| Echocardiogram/MUGA <sup>f</sup> | X | | | | X | X | | X | | X | | X | |
| Confirm Contraceptive Measures <sup>g</sup> | X | | | | | | | | | | | | |
| Study Drug Injection/ Injection<br>Site Reaction Monitoring <sup>h</sup> | | X | X | X | | X | | X | | X | | | |
| Dispensation of Subject Diary<br>Card <sup>i</sup> | | X | X | X | | X | | X | | X | | | |

| Assessment | Screening | (Every | | (Eve | End<br>of<br>Study | Post<br>Study<br>Follow<br>Up | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | Day<br>-28 to -1 | Baseline/ | 3 | 6 | 9 | 18 | 21 | 30 | 33 | 42 | 45 | | |
| Review of Subject Diary Cardi | | | X | X | X | | X | | X | | X | X | |
| Telephone Contact 72 Hours Post<br>Injection | | X | X | X | | X | | X | | X | | | |
| Tumor Imaging <sup>j</sup> | X | | | | X | X | | X | | X | | X | |
| Pregnancy Test <sup>k</sup> | $X^b$ | X <sup>b</sup> | X | X | | X | | X | | X | | X | |
| Urinalysis | X | | | | X | | | X | | | | X | |
| Chemistry Panel | X <sup>b</sup> | X <sup>b</sup> | X | X | X | X | | X | | X | | X | |
| CBC, Differential, Platelets | X <sup>b</sup> | X <sup>b</sup> | X | X | X | X | | X | | X | | X | |
| Coagulation | X | | | | X | | | | | X | | X | |
| Serum Virology (HIV, HBV, HCV) <sup>1</sup> | X | | | | | | | | | | | | |
| Adverse Events | | X | X | X | X | X | X | X | X | X | X | X | |
| Exploratory Immune Analysis | | X | X | X | X | X | X | X | X | X | X | | |
| Exploratory Genomics,<br>Transcriptomics, and Proteomics<br>Molecular Analysis | X | | | | | | | | | | | | |
| Telephone Follow Up <sup>m</sup> | | | | | | | | | | | | | X |

### APPENDIX 2. SPONSOR SIGNATURE

| Study Title: | Phase I Study of Ad5 [E1-, E2b-]-HER2/neu Vaccine (ETBX-021) in Subjects with Unresectable Locally Advanced or Metastatic HER2-Low-Expressing (IHC 1+/2+) Breast Cancer |
|---|---|
| Study Number: | CMS-005, Amendment 2 |
| Final Date: | 25 May 2016 |

This clinical study protocol was subject to critical review and has been approved by the Sponsor. The following personnel contributed to writing and/or approving this protocol:

Date: \_5/25 | 16

Signed:

Wayne R. Godfrey, MD Chief Medical Officer Medical and Safety Monitor NantBioScience, Inc.

# PROTOCOL NUMBER QUILT-3.013 (CMS-005) PHASE 1 STUDY OF AD5 [E1-, E2B-]-HER2/NEU VACCINE (ETBX-021) IN SUBJECTS WITH UNRESECTABLE LOCALLY ADVANCED OR METASTATIC HER2-EXPRESSING (IHC 1+/2+/3+) CANCER

| IND Number: | 016,871 |
|---|---|
| Clinical Study Sponsor: | NantBioScience, Inc. |
| Sponsor Contact:<br>(For medical questions/emergencies) | John H. Lee, MD Senior Vice President Adult Medical Affairs, NantKwest Inc. 9920 Jefferson Blvd Culver City, CA 90232 Email: John.Lee@Nantkwest.com Cell Phone: +1-605-610-6391 |
| Sponsor Contact:<br>(For study administration, operations, and execution questions) | Jim Farmer Senior Director, Clinical Operations NantKwest, Inc Email: Jim.Farmer@Nantkwest.com Office Phone: 310-853-7522 |
| SAE Reporting: | Submit SAE Reports to one of the following:<br>SAE Email: SAE.Reporting@NantBio.com<br>Fax: 800-853-3497 |

| Protocol Version | Date |
|-----------------------------------------------|------------------|
| Original Protocol CMS-005 | 26 February 2016 |
| Protocol CMS-005 Amendment 1 | 20 April 2016 |
| Protocol CMS-005 Amendment 2 | 25 May 2016 |
| Protocol QUILT-3.013 (CMS-005)<br>Amendment 3 | 22 February 2018 |

### PROTOCOL SYNOPSIS

### Name of Sponsor/Company:

NantBioScience, Inc.

### Name of Investigational Product:

Ad5 [E1-, E2b-]-HER2/neu Vaccine, Suspension for Injection (ETBX-021)

### **Name of Active Ingredient:**

Ad5 [E1-, E2b-]-HER2/neu

### Title of Study:

Phase 1 Study of Ad5 [E1-, E2b-]-HER2/neu Vaccine (ETBX-021) in Subjects with Unresectable Locally Advanced or Metastatic HER2-Expressing (IHC 1+/2+/3+) Cancer

### **Study Number:**

QUILT-3.013 (formerly CMS-005)

### **Study Phase:**

Phase 1

### **Primary Objectives:**

• Determine the overall safety and recommended phase 2 dose of ETBX-021 when administered subcutaneously (SC) every 3 weeks for three injections followed by three booster injections at 3-month intervals to subjects with HER2-expressing cancer.

### **Secondary Objectives:**

• Make preliminary assessments of objective response rate (ORR), disease control rate (DCR), duration of response, progression-free survival (PFS), and overall survival (OS) in subjects with HER2-expressing cancer treated with ETBX-021.

### **Exploratory Objectives:**

Evaluate the immunogenicity of ETBX-021 and determine the genomic and proteomic profile
of subjects' tumors to identify gene mutations, gene amplifications, RNA-expression levels,
and protein-expression levels. Correlations between genomic/proteomic profiles and efficacy
outcomes will be assessed.

### **Primary Endpoints:**

- Dose-limiting toxicities (DLTs) and maximum tolerated dose (MTD) or highest tested dose (HTD).
- Treatment-emergent adverse event (AEs) and serious adverse events (SAEs).
- Clinically significant changes in safety laboratory tests, physical examinations, electrocardiograms (ECGs), left ventricular ejection fraction (LVEF), and vital signs.

### **Secondary Endpoints:**

- ORR (confirmed complete or partial response) according to the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
- DCR (confirmed response or stable disease lasting for at least 6 months).
- Duration of response.
- PFS.
- OS.

### **Exploratory Endpoints:**

- Immunogenicity of ETBX-021 by flow cytometric analysis of T-cell frequency, activation status, cytokine profiles, and antibody levels.
- Genetic and proteomic profiling and correlations with efficacy.

### **Study Design:**

This is a phase 1 trial in subjects with unresectable locally advanced or metastatic HER2-expressing (IHC 1+, 2+, or 3+) cancer. The study will be conducted in two parts: the first part will involve dose escalation using a 3 + 3 design, and the second part will involve the expansion of the MTD or HTD to further evaluate safety, preliminary efficacy, and immunogenicity. In the first part, 3 to 6 subjects will be sequentially enrolled starting at dose cohort 1. Subjects will be assessed for dose-limiting toxicities (DLTs).

- Cohort 1:  $5 \times 10^{10}$  virus particles (VP).
- Cohort 2:  $5 \times 10^{11}$  VP.
- If needed, dose de-escalation cohort (cohort -1):  $5 \times 10^9$  VP.

Dose expansion will occur when the MTD or HTD has been determined. An additional 12 subjects will be enrolled in the dose expansion component of the trial, for a total of 18 subjects at the MTD or HTD.

### **Enrollment (planned):**

Up to 30 subjects will be enrolled in the study. In the dose escalation component, 3 to 6 subjects will be sequentially enrolled starting at cohort 1. In the dose expansion component (ie, once the MTD or HTD has been identified), an additional 12 subjects will be enrolled for a total of 18 subjects in the MTD/HTD cohort to obtain further safety, preliminary efficacy, and immunogenicity data.

### Diagnosis and Main Criteria for Inclusion:

Subjects must have histologically confirmed unresectable locally advanced or metastatic cancer that expresses HER2 (IHC 1+, 2+, or 3+).

### **Investigational Product, Dosage, and Mode of Administration:**

ETBX-021 ( $5 \times 10^9$ ,  $5 \times 10^{10}$ , or  $5 \times 10^{11}$  VP in 1.0 mL) will be administered by SC injection every 3 weeks for 3 injections, followed by 3 booster injections at 3-month intervals.

### **Duration of Treatment:**

Subjects will receive treatment for up to 42 weeks (injections at 0, 3, and 6 weeks with booster injections at 18, 30, and 42 weeks) or until they experience progressive disease or unacceptable toxicity, withdraw consent, or if the Investigator feels it is no longer in their best interest to continue treatment.

### Reference Therapy, Dosage, and Mode of Administration:

Not applicable.

### **Criteria for Evaluation:**

**Safety:** Safety endpoints include assessments of DLT, MTD or HTD, treatment-emergent AEs, SAEs, and clinically significant changes in safety laboratory tests, physical examinations, ECGs, LVEF, and vital signs. Toxicities will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03.

**Efficacy:** Tumor response (ORR and DCR) will be evaluated according to RECIST Version 1.1; duration of response, PFS, and OS will also be evaluated.

**Exploratory Immune Analysis:** Immune responses will be detected and quantified in flow cytometry-based and serum assays.

Clinical Trial Protocol: QUILT-3.013 (CMS-005) Amendment 3

Exploratory Molecular Profiling, Analysis, and Rationale: Genomic sequencing of tumor cells from tissue relative to non-tumor cells from whole blood will be profiled to identify the genomic variances that may contribute to response or disease progression and provide an understanding of molecular abnormalities. RNA sequencing will be conducted to provide expression data and give relevance to DNA mutations. Quantitative proteomics analysis will be conducted to determine the exact amounts of specific proteins and to confirm expression of genes that are correlative of response to vaccine immunotherapy and disease progression. All genomic, transcriptomic, and proteomic molecular analyses will be retrospective and exploratory.

### **Statistical Methods:**

The rate of DLTs and the MTD or HTD will be assessed. Overall safety will be assessed by descriptive analyses using tabulated frequencies of AEs by grade using CTCAE Version 4.03 within dose cohorts and for the overall study population in terms of treatment-emergent AEs, SAEs, and clinically significant changes in safety laboratory tests, physical examinations, ECGs, LVEF, and vital signs. ORR and DCR will be evaluated according to RECIST Version 1.1 by dose cohort and overall; duration of response will also be evaluated. PFS and OS will be analyzed using Kaplan-Meier methods by dose cohort and overall.

Figure 1: Study Design and Treatment Schema



**Table 3:** Time and Events Schedule

ETBX-021

| Assessment | Screening | T<br>(Every | | (Evei | End<br>of<br>Study | Post<br>Study<br>Follow<br>Up | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | Day<br>-28 to -1 | Baseline/ | 3 | 6 | 9 | 18 | 21 | 30 | 33 | 42 | 45 | |
| Clinic Visit | X | X | X | X | X | X | X | X | X | X | X | X |
| Informed Consent | X | | | | | | | | | | | |
| Inclusion/Exclusion | X | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | |
| Physical Examination, Height <sup>a</sup> , Weight, ECOG | $X^{b}$ | $X^b$ | X | X | X | X | | X | | X | | X |
| Medical History <sup>c</sup> | X | X | | | | | | | | | | |
| Confirm HER2 Expression <sup>d</sup> | X | | | | | | | | | | | |
| Concomitant Medications | X | X | X | X | X | X | | X | | X | | X |
| Vital Signs <sup>e</sup> | X | X | X | X | X | X | | X | | X | | X |
| 12-Lead ECG | X | | | | X | X | | X | | X | | X |
| Echocardiogram/MUGA <sup>f</sup> | X | | | | X | X | | X | | X | | X |
| Confirm Contraceptive Measures <sup>g</sup> | X | | | | | | | | | | | |
| Study Drug Injection/ Injection<br>Site Reaction Monitoring <sup>h</sup> | | X | X | X | | X | | X | | X | | |
| Dispensation of Subject Diary<br>Card <sup>i</sup> | | X | X | X | | X | | X | | X | | |

| Assessment | Screening | T<br>(Every : | | (Eve | End<br>of<br>Study | Post<br>Study<br>Follow<br>Up | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | Day<br>-28 to -1 | Baseline/ | 3 | 6 | 9 | 18 | 21 | 30 | 33 | 42 | 45 | | |
| Review of Subject Diary Card <sup>i</sup> | | | X | X | X | | X | | X | | X | X | |
| Telephone Contact 72 Hours Post<br>Injection | | X | X | X | | X | | X | | X | | | |
| Tumor Imaging <sup>j</sup> | X | | | | X | X | | X | | X | | X | |
| Pregnancy Test <sup>k</sup> | $X^{b}$ | X <sup>b</sup> | X | X | | X | | X | | X | | X | |
| Urinalysis | X | | | | X | | | X | | | | X | |
| Chemistry Panel | X <sup>b</sup> | X <sup>b</sup> | X | X | X | X | | X | | X | | X | |
| CBC, Differential, Platelets | X <sup>b</sup> | X <sup>b</sup> | X | X | X | X | | X | | X | | X | |
| Coagulation | X | | | | X | | | | | X | | X | |
| Serum Virology (HIV, HBV, HCV) <sup>1</sup> | X | | | | | | | | | | | | |
| Adverse Events | | X | X | X | X | X | X | X | X | X | X | X | |
| Exploratory Immune Analysis | | X | X | X | X | X | X | X | X | X | X | | |
| Exploratory Genomics,<br>Transcriptomics, and Proteomics<br>Molecular Analysis | X | | | | | | | | | | | | |
| Telephone Follow Up <sup>m</sup> | | | | | | | | | | | | | X |

Date: Feb 22 20/8

### APPENDIX 2. SPONSOR SIGNATURE

| Study Title: | Phase 1 Study of Ad5 [E1-, E2b-]-HER2/neu Vaccine (ETBX-021) in Subjects with Unresectable Locally Advanced or Metastatic HER2-expressing (IHC 1+/2+/3+) Cancer |
|---|---|
| Study Number: | QUILT-3.013 (CMS-005), Amendment 3 |
| Final Date: | 22 February 2018 |

This clinical study protocol was subject to critical review and has been approved by NantBioScience, Inc. The following personnel contributed to writing and/or approving this

protocol:

Signed:

John H. Lee, MD

Senior Vice President Adult Medical Affairs,

NantKwest Inc. 9920 Jefferson Blvd Culver City, CA 90232

Email: John.Lee@Nantkwest.com

Cell Phone: +1-605-610-6391

# PROTOCOL NUMBER QUILT-3.013 (CMS-005) PHASE 1 STUDY OF AD5 [E1-, E2B-]-HER2/NEU VACCINE (ETBX-021) IN SUBJECTS WITH UNRESECTABLE LOCALLY ADVANCED OR METASTATIC HER2-EXPRESSING (IHC 1+/2+/3+) CANCER

| IND Number: | 016,871 |
|---|---|
| Clinical Study Sponsor: | NantBio, Inc. |
| Sponsor Contact:<br>(For medical questions/emergencies) | John H. Lee, MD Senior Vice President Adult Medical Affairs, NantKwest Inc. 9920 Jefferson Blvd Culver City, CA 90232 Email: John.Lee@Nantkwest.com Cell Phone: +1-605-610-6391 |
| Sponsor Contact:<br>(For study administration, operations, and execution questions) | Jim Farmer Senior Director, Clinical Operations NantKwest, Inc Email: Jim.Farmer@Nantkwest.com Office Phone: 310-853-7522 |
| SAE Reporting: | Submit SAE Reports to one of the following:<br>SAE Email: SAE.Reporting@NantBio.com<br>Fax: 800-853-3497 |

| Protocol Version | Date |
|--------------------------------|------------------|
| Original Protocol CMS-005 | 26 February 2016 |
| Protocol CMS-005 Amendment 1 | 20 April 2016 |
| Protocol CMS-005 Amendment 2 | 25 May 2016 |
| Protocol QUILT-3.013 (CMS-005) | 22 February 2018 |
| Amendment 3 | |
| Protocol QUILT-3.013 (CMS-005) | 1 May 2018 |
| Amendment 4 | |

ETBX-021 NantBio, Inc.

### PROTOCOL SYNOPSIS

### Name of Sponsor/Company:

NantBio, Inc.

### **Name of Investigational Product:**

Ad5 [E1-, E2b-]-HER2/neu Vaccine, Suspension for Injection (ETBX-021)

### **Name of Active Ingredient:**

Ad5 [E1-, E2b-]-HER2/neu

### Title of Study:

Phase 1 Study of Ad5 [E1-, E2b-]-HER2/neu Vaccine (ETBX-021) in Subjects with Unresectable Locally Advanced or Metastatic HER2-Expressing (IHC 1+/2+/3+) Cancer

### **Study Number:**

QUILT-3.013 (formerly CMS-005)

### **Study Phase:**

Phase 1

### **Primary Objectives:**

• Determine the overall safety and recommended phase 2 dose of ETBX-021 when administered subcutaneously (SC) every 3 weeks for three injections followed by three booster injections at 3-month intervals to subjects with HER2-expressing cancer.

### **Secondary Objectives:**

 Make preliminary assessments of objective response rate (ORR), disease control rate (DCR), duration of response, progression-free survival (PFS), and overall survival (OS) in subjects with HER2-expressing cancer treated with ETBX-021.

### **Exploratory Objectives:**

Evaluate the immunogenicity of ETBX-021 and determine the genomic and proteomic profile
of subjects' tumors to identify gene mutations, gene amplifications, RNA-expression levels,
and protein-expression levels. Correlations between genomic/proteomic profiles and efficacy
outcomes will be assessed.

### **Primary Endpoints:**

- Dose-limiting toxicities (DLTs) and maximum tolerated dose (MTD) or highest tested dose (HTD).
- Treatment-emergent adverse event (AEs) and serious adverse events (SAEs).
- Clinically significant changes in safety laboratory tests, physical examinations, electrocardiograms (ECGs), left ventricular ejection fraction (LVEF), and vital signs.

### **Secondary Endpoints:**

- ORR (confirmed complete or partial response) according to the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
- DCR (confirmed response or stable disease lasting for at least 6 months).
- Duration of response.
- PFS.
- OS.

ETBX-021 NantBio, Inc.

### **Exploratory Endpoints:**

- Immunogenicity of ETBX-021 by flow cytometric analysis of T-cell frequency, activation status, cytokine profiles, and antibody levels.
- Genetic and proteomic profiling and correlations with efficacy.

### **Study Design:**

This is a phase 1 trial in subjects with unresectable locally advanced or metastatic HER2-expressing (IHC 1+, 2+, or 3+) cancer. The study will be conducted in two parts: the first part will involve dose escalation using a 3 + 3 design, and the second part will involve the expansion of the MTD or HTD to further evaluate safety, preliminary efficacy, and immunogenicity. In the first part, 3 to 6 subjects will be sequentially enrolled starting at dose cohort 1. Subjects will be assessed for dose-limiting toxicities (DLTs).

- Cohort 1:  $5 \times 10^{10}$  virus particles (VP).
- Cohort 2:  $5 \times 10^{11}$  VP.
- If needed, dose de-escalation cohort (cohort -1):  $5 \times 10^9$  VP.

Dose expansion will occur when the MTD or HTD has been determined. An additional 12 subjects will be enrolled in the dose expansion component of the trial, for a total of 18 subjects at the MTD or HTD.

### **Enrollment (planned):**

Up to 30 subjects will be enrolled in the study. In the dose escalation component, 3 to 6 subjects will be sequentially enrolled starting at cohort 1. In the dose expansion component (ie, once the MTD or HTD has been identified), an additional 12 subjects will be enrolled for a total of 18 subjects in the MTD/HTD cohort to obtain further safety, preliminary efficacy, and immunogenicity data.

### Diagnosis and Main Criteria for Inclusion:

Subjects must have histologically confirmed unresectable locally advanced or metastatic cancer that expresses HER2 (IHC 1+, 2+, or 3+). For malignancies other than breast and gastrointestinal, HER2 expression must be confirmed by a validated in situ hybridization (ISH) assay with results considered positive of HER2 amplification by ASCO/CAP HER2 testing guideline.

### Investigational Product, Dosage, and Mode of Administration:

ETBX-021 ( $5 \times 10^9$ ,  $5 \times 10^{10}$ , or  $5 \times 10^{11}$  VP in 1.0 mL) will be administered by SC injection every 3 weeks for 3 injections, followed by 3 booster injections at 3-month intervals.

### **Duration of Treatment:**

Subjects will receive treatment for up to 42 weeks (injections at 0, 3, and 6 weeks with booster injections at 18, 30, and 42 weeks) or until they experience progressive disease or unacceptable toxicity, withdraw consent, or if the Investigator feels it is no longer in their best interest to continue treatment.

### Reference Therapy, Dosage, and Mode of Administration:

Not applicable.

### **Criteria for Evaluation:**

**Safety:** Safety endpoints include assessments of DLT, MTD or HTD, treatment-emergent AEs, SAEs, and clinically significant changes in safety laboratory tests, physical examinations, ECGs, LVEF, and vital signs. Toxicities will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03.

**Efficacy:** Tumor response (ORR and DCR) will be evaluated according to RECIST Version 1.1; duration of response, PFS, and OS will also be evaluated.

ETBX-021 NantBio, Inc.

**Exploratory Immune Analysis:** Immune responses will be detected and quantified in flow cytometrybased and serum assays.

Exploratory Molecular Profiling, Analysis, and Rationale: Genomic sequencing of tumor cells from tissue relative to non-tumor cells from whole blood will be profiled to identify the genomic variances that may contribute to response or disease progression and provide an understanding of molecular abnormalities. RNA sequencing will be conducted to provide expression data and give relevance to DNA mutations. Quantitative proteomics analysis will be conducted to determine the exact amounts of specific proteins and to confirm expression of genes that are correlative of response to vaccine immunotherapy and disease progression. All genomic, transcriptomic, and proteomic molecular analyses will be retrospective and exploratory.

### **Statistical Methods:**

The rate of DLTs and the MTD or HTD will be assessed. Overall safety will be assessed by descriptive analyses using tabulated frequencies of AEs by grade using CTCAE Version 4.03 within dose cohorts and for the overall study population in terms of treatment-emergent AEs, SAEs, and clinically significant changes in safety laboratory tests, physical examinations, ECGs, LVEF, and vital signs. ORR and DCR will be evaluated according to RECIST Version 1.1 by dose cohort and overall: duration of response will also be evaluated. PFS and OS will be analyzed using Kaplan-Meier methods by dose cohort and overall.

Figure 1: Study Design and Treatment Schema



**Table 3:** Time and Events Schedule

| Assessment | Screening Treatment Boosters (Every 3-Week Dosing) (Every 3-Month Dosing) | | | | | | | | | End<br>of<br>Study | Post<br>Study<br>Follow<br>Up | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | Day<br>-28 to -1 | Baseline/ | 3 | 6 | 9 | 18 | 21 | 30 | 33 | 42 | 45 | |
| Clinic Visit | X | X | X | X | X | X | X | X | X | X | X | X |
| Informed Consent | X | | | | | | | | | | | |
| Inclusion/Exclusion | X | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | |
| Physical Examination, Height <sup>a</sup> , Weight, ECOG | $X^b$ | $X^b$ | X | X | X | X | | X | | X | | X |
| Medical History <sup>c</sup> | X | X | | | | | | | | | | |
| Confirm HER2 Expression <sup>d</sup> | X | | | | | | | | | | | |
| Concomitant Medications | X | X | X | X | X | X | | X | | X | | X |
| Vital Signs <sup>e</sup> | X | X | X | X | X | X | | X | | X | | X |
| 12-Lead ECG | X | | | | X | X | | X | | X | | X |
| Echocardiogram/MUGA <sup>f</sup> | X | | | | X | X | | X | | X | | X |
| Confirm Contraceptive Measures <sup>g</sup> | X | | | | | | | | | | | |
| Study Drug Injection/ Injection<br>Site Reaction Monitoring <sup>h</sup> | | X | X | X | | X | | X | | X | | |
| Dispensation of Subject Diary<br>Card <sup>i</sup> | | X | X | X | | X | | X | | X | | |

| Assessment | Screening | | Treatment Boosters (Every 3-Week Dosing) (Every 3-Month Dosing) | | | | | | | | End<br>of<br>Study | Post<br>Study<br>Follow<br>Up | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | Day -28 to -1 | Baseline/ | 3 | 6 | 9 | 18 | 21 | 30 | 33 | 42 | 45 | | |
| Review of Subject Diary Card <sup>i</sup> | | | X | X | X | | X | | X | | X | X | |
| Telephone Contact 72 Hours Post<br>Injection | | X | X | X | | X | | X | | X | | | |
| Tumor Imaging <sup>j</sup> | X | | | | X | X | | X | | X | | X | |
| Pregnancy Test <sup>k</sup> | X <sup>b</sup> | X <sup>b</sup> | X | X | | X | | X | | X | | X | |
| Urinalysis | X | | | | X | | | X | | | | X | |
| Chemistry Panel | X <sup>b</sup> | X <sup>b</sup> | X | X | X | X | | X | | X | | X | |
| CBC, Differential, Platelets | X <sup>b</sup> | X <sup>b</sup> | X | X | X | X | | X | | X | | X | |
| Coagulation | X | | | | X | | | | | X | | X | |
| Serum Virology (HIV, HBV, HCV) <sup>1</sup> | X | | | | | | | | | | | | |
| Adverse Events | | X | X | X | X | X | X | X | X | X | X | X | |
| Exploratory Immune Analysis | | X | X | X | X | X | X | X | X | X | X | | |
| Exploratory Genomics,<br>Transcriptomics, and Proteomics<br>Molecular Analysis | X | | | | | | | | | | | | |
| Telephone Follow Up <sup>m</sup> | | | | | | | | | | | | | X |

### APPENDIX 2. SPONSOR SIGNATURE

| Study Title: | Phase 1 Study of Ad5 [E1-, E2b-]-HER2/neu Vaccine (ETBX-021) in Subjects with Unresectable Locally Advanced or Metastatic HER2-expressing (IHC 1+/2+/3+) Cancer |
|---|---|
| Study Number: | QUILT-3.013 (CMS-005), Amendment 4 |
| Final Date: | 1 May 2018 |

This clinical study protocol was subject to critical review and has been approved by NantBio, Inc. The following personnel contributed to writing and/or approving this protocol:

Signed:

John H. Lee, MD

Senior Vice President Adult Medical Affairs,

NantKwest Inc.

9920 Jefferson Blvd

Culver City, CA 90232

Email: John.Lee@Nantkwest.com Cell Phone: +1-605-610-6391